CLINICAL TRIAL: NCT01328548
Title: Immune and Genetic Correlates of Response to Zoster Vaccine in the Frail Elderly: a Pilot Study
Brief Title: Zoster Vaccine Response in the Frail Elderly
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-450
Record Dates: First submitted 2011-03-15; First posted 2011-04-04 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Immune System Diseases
Keywords: varicella-zoster virus; vaccine; T-cell; genes; frail elderly; immunosenescence; immune and genetic correlates of response to zoster vaccine in the elderly
MeSH Terms: conditions — Immune System Diseases; Chickenpox | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retained specimens include DNA and blood cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Nursing Home Elderly Cases: Non-ambulatory nursing home residents >= 80 years old will be vaccinated with the zoster vaccine and provide baseline and post-vaccination blood samples. We will assess differences in genotype frequencies between participants with high and low RCF and ELISPOT responses using a candidate gene approach with SNPs (single nucleotide polymorphisms). A case will be considered failure to mount a high response.
  Interventions: Drug: Zostavax
- Nursing Home Elderly Controls: Non-ambulatory nursing home residents >= 80 years old will be vaccinated with the zoster vaccine and provide baseline and post-vaccination blood samples. We will assess differences in genotype frequencies between participants with high and low RCF and ELISPOT responses using a candidate gene approach with SNPs. A control will be a participant who mounted an adequate response as defined in primary outcomes.
  Interventions: Drug: Zostavax
- Community dwelling seniors: Community dwelling seniors ages 60-75 will be enrolled as a control group for the laboratory testing. They will be vaccinated and will provide pre- and post-vaccination blood. If nursing home residents do not show a response it is important to know that it is not a failure of the laboratory's measurement of immunogenicity.
  Interventions: Drug: Zostavax

INTERVENTIONS:
Drug: Zostavax
  Other Names: Zoster vaccine

SUMMARY:
This study is being done to evaluate the zoster vaccine response in the nursing home elderly (80 years or older). As the immune system ages, the response to vaccines is not always as strong as in younger people. Previous zoster vaccine studies have excluded nursing home residents so the vaccine effect in this population is not known. Furthermore, the immune and genetic reasons as to why the vaccine works well in some people but not in others are also unknown. The goal of this study is to evaluate why some immune systems respond well to the vaccine and why others do not.

DETAILED DESCRIPTION:
Deleterious changes in immunity that occur with aging are known as immunosenescence. Such changes, particularly in adaptive immunity, may lead to an impaired vaccine response in the elderly. Characterizing the immune determinants and the genetic basis for vaccine response in the frail elderly is a practical approach to better our understanding of immunosenescence. Data on genetic determinants to immunization are sparse, furthermore, to the best of our knowledge, none exist in the elderly. In this pilot study, we propose studying the immune response to the herpes zoster vaccine and the underlying genetic determinants of the immune response in elderly residents of nursing homes.

The three specific aims of this study are to generate data in order to 1) assess the T-cell response to the varicella-zoster virus (VZV) vaccine in the frail elderly; 2) assess whether immune (T-cell) phenotypes are associated with a response; 3) test the association between immune response genotype sets and T-cell response. We hypothesize that response to the VZV vaccine in elderly nonambulatory nursing home residents is a function of characteristic T-cell immune phenotypes prior to vaccination and that there are immune genetic polymorphisms associated with the response. This study will allow us to generate preliminary data and establish feasibility in order to address these questions fully in a larger population in a subsequent grant application.

ELIGIBILITY:
Inclusion Criteria:

* nursing home resident
* greater than or equal to 80 years old
* non-ambulatory

Exclusion Criteria:

* less than 80 years old
* ambulatory
* taking immunosuppressive medication
* history of primary or acquired immuno-deficiency states including leukemia, other malignant neoplasms affecting the bone marrow or lymphatic system, and AIDS
* active untreated tuberculosis
* previous receipt of varicella vaccine
* residents expected to expire within 30 days, in the opinion of the most responsible physician
* residents planning to move nursing homes within the year
* temporary residents

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly, non-ambulatory residents of nursing homes.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark B. Loeb, FRCPC,MD,MSc, Principal Investigator — McMaster University
Locations (1):
- Macassa Lodge, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Lelic A, Verschoor CP, Lau VW, Parsons R, Evelegh C, Bowdish DM, Bramson JL, Loeb MB. Immunogenicity of Varicella Vaccine and Immunologic Predictors of Response in a Cohort of Elderly Nursing Home Residents. J Infect Dis. 2016 Dec 15;214(12):1905-1910. doi: 10.1093/infdis/jiw462. Epub 2016 Oct 5. PMID 27707807

RESULTS

PARTICIPANT FLOW:
Groups:
- Nursing Home Vaccine Group: Nursing home residents >= 80 years vaccinated with the ZOSTAVAX zoster vaccine
- Community Control Vaccine Group: Community dwelling seniors ages 60-75 years vaccinated with the Zostavax zoster vaccine
Period: Overall Study
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Started | 191 | 50
Completed | 187 | 50
Not Completed | 4 | 0
Not completed — Death | 3 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group | Total
Number analyzed (Participants) | 191 | 50 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 15 | 15
  >=65 years | 191 | 35 | 226
Age, Continuous [Mean (Standard Deviation); unit: Years] | 89.0 (4.69) | 67.3 (4.34) | 84.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 32 | 186
  Male | 37 | 18 | 55
Region of Enrollment [Number; unit: Participants]
  Canada | 191 | 50 | 241

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in T-cell Response to the VZV Vaccine in the Frail Elderly
Description: As the primary phenotype, we will compare change in Enzyme-linked immunosorbent spot (ELISPOT) from baseline (i.e., pre and post vaccination). A high baseline T cell response will be defined as ELISPOT = >50 spots and a low baseline response will be ELISPOT = <10 spots.
Time Frame: 6 weeks
Population: IFN-gamma T cell ELISpot assay (sfu) against VZV taken prior to vaccination and 6 weeks post vaccination
Measure: Mean (Standard Deviation); unit: Spot Forming Units per 10^6 PBMC
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Number analyzed (Participants) | 187 | 50
Spot Forming Units per 10^6 PBMC
  Pre-vaccine IFN-gamma T cell ELISpot assay count | 50.17 (54.84) | 78.17 (65.37)
  Post- vaccine IFN-gamma T cell ELISpot assay count | 83.22 (72.56) | 120.56 (76.87)

2. Primary Outcome: Assessment of Immune Parameters Compatible With Inflammaging: CD4+/CD8+ Ratio
Description: Characterization of T-cell populations will be conducted on whole blood using multi-parametric flow cytometry prior to immunization to characterize the immunological function of circulating T-cells in the nursing home vaccine group.
Time Frame: Baseline
Population: Predictor variables were assessed only among the frail elderly, the community control group served as a control for immunogenicity only.
Measure: Mean (Standard Deviation); unit: T-cell ratio
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Number analyzed (Participants) | 186 | 0
T-cell ratio | 3.06 (2.38) |

3. Primary Outcome: Assessment of Immune Parameters Compatible With Inflammaging: High T Regulatory Cells
Description: as for outcome 2
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of peripheral blood mononuclear cell
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Number analyzed (Participants) | 186 | 0
% of peripheral blood mononuclear cell | 2.23 (1.00) |

4. Other Pre Specified Outcome: Assessment of Immune Parameters Compatible With Inflammaging: TEMRA Cells
Description: Characterization of Tcell populations will be conducted on whole blood using multiparametric flow cytometry prior to immunization to characterize the immunological function of circulating Tcells in each participant.
Time Frame: Baseline
Population: Data not collected.
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Assessment of Immune Parameters Compatible With Inflammaging: High CD8+CD28CD45RA+T Cells
Description: as for outcome 4
Time Frame: Baseline
Population: Data not collected.
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Testing 150 Candidate Immune Response Genes for SNP Analysis
Description: These will include Tolllike receptors, cytokines, chemokines, chemokine receptors, interferons and interferon receptors. Tolllike receptors: TLR1TLR9 Cytokines: ILI1A, ILI1B, IL1RN, IL4, IL5, IL12B, IL13, CSF2 Chemokines: CCL1CCL3, CCL3L1, CCL4CCL8, CCL11, CCL13, CCL15CCL28, CXCL1CXCL14, CXCL16, CX3CL1 Chemokine receptors: CCR1CCR10, CXCR1CXCR6, CX3CR1, XCR1XCR2 Interferons: IFNA1IFNA2, IFNA4IFNA8, IFNA10, IFNA13, IFNA14, IFNA16IFNA17, IFNA21, IFNB1, IFNB3, IFNG, IFNK, IFNW1 Interferon receptors: IFNAR1, IFNAR2, IFNGR1, IFNGR2
Time Frame: Baseline
Population: Genotyping was not conducted because of insufficient resources.
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Assessment of Immune Parameters Compatible With Inflammaging: CD4 Cell Frequency
Description: as for outcome 2
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of peripheral blood mononuclear cell
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Number analyzed (Participants) | 186 | 0
% of peripheral blood mononuclear cell | 65.24 (15.41) |

ADVERSE EVENTS:
Arm/Group | Nursing Home Vaccine Group | Community Control Vaccine Group
Serious Adverse Events (participants affected / at risk) | 3/191 | 0/50
Other Adverse Events (participants affected / at risk) | 23/191 | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nursing Home Vaccine Group (N=191) | Community Control Vaccine Group (N=50)
Pre-existing fragile health and advanced age (General disorders) | 1 (1) | 0 (0) — Non-vaccine related death
Progressive renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Non-vaccine related death
Advanced age and medical issues (Parkinson's disease) (Nervous system disorders) | 1 (1) | 0 (0) — Non-vaccine related death
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nursing Home Vaccine Group (N=191) | Community Control Vaccine Group (N=50)
Cough (General disorders) | 4 (4) | 0 (0)
Fall (General disorders) | 3 (3) | 0 (0)
Lethargy (General disorders) | 5 (5) | 0 (0)
Emesis/Nausea (General disorders) | 5 (5) | 0 (0)
Pain/Soreness in arm (General disorders) | 3 (3) | 2 (2)
Redness/Swelling in arm (General disorders) | 4 (4) | 9 (9)
Headache (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No